CLINICAL TRIAL: NCT00255970
Title: Regenerative Therapy for Vertical Defects Comparing Demineralized Freeze Dried Bone Allograft (DFDBA) and Regenafil
Brief Title: Regenafil Versus Demineralized Freeze Dried Bone Allograft (DFDBA) for Periodontal Defects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor, Regeneration Technologies, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RegenF052005
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Results first posted 2011-08-05 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Periodontal Diseases
Keywords: Periodontal Treatment of Intraosseous Vertical Defects
MeSH Terms: conditions — Periodontal Diseases | interventions — Grafton demineralized bone matrix gel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regenafil graft (Experimental): Regenafil
  Interventions: Device: Regenafil
- DFDBA (Active Comparator): Demineralized Freeze Dried Bone Allograft
  Interventions: Other: DFDBA; Device: Regenafil

INTERVENTIONS:
Other: DFDBA — Demineralized Freeze Dried Allograft bone
  Other Names: Demineralized Bone Matrix
  Arms: DFDBA
Device: Regenafil — Demineralized Freeze Dried Bone in a porcine gel carrier
  Other Names: Demineralized Freeze Dried Bone Allograft

SUMMARY:
The purpose of this research study was to determine whether treatment with the bone grafting material Regenafil was as effective as the standard treatment using demineralized freeze dried bone allograft (DFDBA). Regenafil is demineralized freeze dried bone in a special gel form.

DETAILED DESCRIPTION:
To compare the regenerative effects of a demineralized freeze dried bone allograft (DFDBA) particulate in a biologic thermoplastic carrier (Regenafil) to the standard of care. To compare the regenerative effects of a demineralized freeze dried bone allograft (DFDBA) particulate in the treatment of intraosseous vertical defects following six months of healing. This was accomplished by evaluating clinical parameters including probing depth, attachment level and bleeding upon probing, using attachment level as the primary outcome variable.

Treatment of the vertical osseous defect is a challenging problem in periodontics. There are many treatment options including:

1. open flap debridement;
2. osseous graft alone;
3. membrane alone;
4. or membrane plus an osseous graft.

Choice of treatment may depend on the defect depth and configuration. A shallow, narrow 3 wall defect may respond well to open flap debridement while a deep 2 wall defect may need regenerative therapy such as an osseous graft, a membrane or combined membrane and graft treatment. Studies of vertical defect therapy with defects about 4 mm or greater show that similar percent defect fill results are obtained with regenerative therapies. Open flap debridement produces substantially less percent defect fill.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to their participation.
2. Be an adult age 18 and older.
3. Have at least a 4 mm open vertical osseous defect depth on one tooth, visible on a radiograph and with a probing depth ≥ 5 mm.
4. Have osseous defects that are either wide 3-wall, or combination defects.

Exclusion Criteria:

1. Have debilitating systemic diseases, or diseases that affect the periodontium.
2. Have a known allergy to any of the materials that will be used in the study:

   * non-steroidal anti-inflammatory drugs (NSAIDs)
   * chlorhexidine digluconate
   * doxycycline
   * gelatin
3. Need prophylactic antibiotics.
4. Have a vertical osseous defect that is related to a furcation area.
5. Smoke more than 1 pack per day.
6. Have endodontically treated teeth or endodontic lesions at study sites.
7. Have 1-wall defects.
8. Have poor oral hygiene.
9. Have anterior fillings (Note: if a subject presents with anterior fillings, it will be at the discretion of the principal investigator as to whether they should be accepted into the study.)
10. Be pregnant as evidenced by a positive urine pregnancy test taken at both the screening and baseline visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville; Steven Blanchard, DDS, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University School of Dentistry, Indianapolis, Indiana
  - University of Louisville School of Dentistry, Louisville, Kentucky

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done through the investigators clinics.
Pre-assignment Details: The was no wash out or run-in events in this study.
Groups:
- Regenafil: Regenafil graft
- Demineralized Freeze Dried Bone Allograft: Demineralized Freeze Dried Bone Allograft (DFDBA)
Period: Overall Study
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft
Started | 21 | 19
Screening Visit | 21 | 19
Final Visit Week 24 | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 4 | 2 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.7) | 51.4 (14) | 51.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 14 | 8 | 22
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Probing Depth
Description: This is the distance, measured in millimeters (mm) from the gingival margin to the maximal penetration of the probe tip. The measures were made at baseline and then at 6 months after treatment.
Time Frame: baseline and then at 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft
Number analyzed (Participants) | 21 | 19
mm | 2.7 (1.1) | 2.4 (1.2)
Statistical Analysis 1: Comparison: Regenafil vs Demineralized Freeze Dried Bone Allograft; This study had been designed as a superiority study. The null hypothesis had been that there would be no significant difference in probing depth between groups at the time points measured; Test type: Superiority or Other; p > .05, ANOVA
Statistical Analysis 2: Comparison: Regenafil vs Demineralized Freeze Dried Bone Allograft; A power analysis, prior to data collection, determined that a minimum of 18 in each arm would be needed for this study; Test type: Superiority or Other; p > 0.05, ANOVA — The power analysis had been computed for a threshold of 0.05 with a power of 0.8

2. Primary Outcome: Clinical Attachment Level
Description: The amount of space between attached periodontal tissues and a fixed point, usually the cementoenamel junction. A measurement used to assess the stability of attachment as part of a periodontal maintenance program.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft
Number analyzed (Participants) | 21 | 19
mm | 5.6 (2.0) | 6.3 (1.9)
Statistical Analysis 1: Comparison: Regenafil vs Demineralized Freeze Dried Bone Allograft; This study had been designed as a superiority study. The a priori power analysis had been designed with an effect size based on historical data. Thus, a minimal sample size of 34 patients would be necessary to determine if there was a true difference between groups, α =.05, power= 0.8. This number was then rounded to 40 patients, 20/ group (DFDBA and Regenafil); Test type: Superiority or Other; p > .05, ANOVA

3. Primary Outcome: Recession
Description: CEJ to gingival margin (GM). GM coronal to the CEJ were scored as a negative number.
Time Frame: 6 months
Population: The number of participants to be analyzed was based on a power analysis, using a threshold of 0.05 with a power of 0.8. The power analysis indicated 18 participants were needed in each arm
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft
Number analyzed (Participants) | 21 | 19
mm | 0.9 (1.1) | 0.9 (1.1)
Statistical Analysis 1: Comparison: Regenafil vs Demineralized Freeze Dried Bone Allograft; The change in recession, measured in mm, had been designed as a superiority study. The a priori power analysis had been designed with an effect size based on historical data. Thus, a minimal sample size of 34 patients would be necessary to determine if there was a true difference between groups, α =.05, power= 0.8. This number was then rounded to 40 patients, 20/ group (DFDBA and Regenafil); Test type: Superiority or Other; p > 0.05, ANOVA

4. Secondary Outcome: Gingival Index
Description: Scores:
  0 Normal gingiva
  1. Mild inflammation
  2. Moderate inflammation
  3. Severe inflammation Gingival units (buccal, lingual, mesiobuccal, distobuccal, mesiolingual, and distolingual) of each tooth were scored 0-3. Scores from the 6 areas of the tooth were added and divided by 6 to give the gingival index for the entire tooth.
Time Frame: 6 months
Population: As stated in the protocol, the power analysis (threshold=0.05, power>0.8) noted 18 subjects would be needed per group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft
Number analyzed (Participants) | 21 | 19
Units on a scale | 0.5 (0.8) | 0.7 (0.8)
Statistical Analysis 1: Comparison: Regenafil vs Demineralized Freeze Dried Bone Allograft; Each gingival unit (buccal, lingual, mesiobuccal, distobuccal, mesiolingual, and distolingual) of the individual tooth will be given a score from 0-3, called the gingival index for the area. The scores from the 6 areas of the tooth are added and divided by 6 to give the gingival index for the tooth; Test type: Superiority or Other; p > 0.05, ANOVA

5. Secondary Outcome: Plaque Index
Description: 0- No plaque
  1. A film of plaque adhering to gingival margin & adjacent area of tooth
  2. Moderate accumulation of soft deposits, visible with the naked eye
  3. Abundance of soft matter Each gingival region of the individual tooth will be scored 0-3 The scores from the 6 areas of the tooth are averaged to give the plaque index for the tooth.
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Categorical index score
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft
Number analyzed (Participants) | 21 | 19
Categorical index score | 0.4 (0.5) | 0.6 (0.5)
Statistical Analysis 1: Comparison: Regenafil vs Demineralized Freeze Dried Bone Allograft; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p > 0.05, ANOVA

6. Secondary Outcome: Bleeding on Probing
Description: The variable measured the presence of bleeding when the osseus defect was probed. The presence and character of gingival bleeding will be determined by gently probing to the base of the pockets.
  0 - No bleeding.
  1 - Bleeding when probing.
Time Frame: 6 months
Population: The a priori power analysis had been designed with an effect size based on historical data. Thus, a minimal sample size of 34 patients would be necessary to determine if there was a true difference between groups, α =.05, power= 0.8. This number was then rounded to 40 patients, 20/ group (DFDBA and Regenafil).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft
Number analyzed (Participants) | 21 | 19
Units on a scale | 0.4 (0.3) | 0.3 (0.3)

7. Secondary Outcome: Mobility Index
Description: Tooth mobility was recorded using Miller's Index:
  1. - up to 1 mm of movement in a horizontal direction
  2. - greater than 1 mm of movement in a horizontal direction
  3. - excessive horizontal movement and vertical movement. Manual evaluation of mobility was carried out clinically using the handles of two instruments to move the teeth buccally and lingually and note their movement.
Time Frame: 6 months
Population: A power analysis, prior to data collection, determined that a minimum of 18 in each arm would be needed for this study. The power analysis had been computed for a threshold of 0.05 with a power of 0.8.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft
Number analyzed (Participants) | 21 | 19
Units on a scale | 0.4 (0.5) | 0.6 (0.5)

ADVERSE EVENTS:
Arm/Group | Regenafil | Demineralized Freeze Dried Bone Allograft
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less